CLINICAL TRIAL: NCT01638624
Title: The Effect of Propofol Infusion on Total Antioxidant Status During Tourniquet-Induced Ischemia-Reperfusion Injury in Total Knee Arthroplasty
Brief Title: The Effect of Propofol Infusion on Total Antioxidant Status During Tourniquet-Induced Ischemia-Reperfusion Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, Consultant MD of Anesthesiology Department, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Diskapi2012
Record Dates: First submitted 2012-07-03; First posted 2012-07-12 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2012-07

CONDITIONS: Total Knee Arthroplasty; Tourniquet-Induced Ischemia-Reperfusion Injury
Keywords: Propofol; antioxidant capacity; total knee arthroplasty; Propofol,antioxidant
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Propofol (Active Comparator): Propofol infusion group: Under spinal anesthesia, a continuous intravenous infusion (2mg/kg/h) of propofol will be use during the operation
  Interventions: Drug: Propofol
- Control group (Placebo Comparator): Placebo group: Under spinal anesthesia, a continuous intravenous infusion of volume-equivalent placebo will use during the operation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propofol — Propofol :Propofol is an anesthetic agent, has structure similar to that of known such as alfa tocopherol.
  Arms: Propofol
Drug: Placebo
  Arms: Control group

SUMMARY:
The release of tourniquet produces reactive oxygen species which can cause injury. Propofol is chemically similar to phenol-based free radical scavengers.

Plasma total antioxidant capacity is a well-established marker of the overall protective effect of antioxidants in body fluids.The aim of the study is to investigate the effects of propofol on ischemia-reperfusion injury in total knee arthroplasty (TKA).

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II physical status
* Unilateral total knee arthroplasty
* Age 18 years to 80 years

Exclusion Criteria:

* Severe central nervous system disorders
* Severe cardiopulmonary,renal,metabolic, or hepatic disease,
* Blood volume deficits,
* Coagulopathy,
* Allergy to local anesthetics,
* Peripheral neuropathies,
* Body mass index > 35,
* History of antioxidant drug use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The perioperative alternation of the venous blood total antioxidant capacity levels of the arms | T1,T2,T3
  T1 : Before the spinal anesthesia performed T2 : At 30th min of tourniquet inflation T3 : At 2nd hours of tourniquet deflation

CONTACTS AND LOCATIONS:
Overall Officials: Derya Özkan, MD, Principal Investigator — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Anesthesiology Clinic; Taylan Akkaya, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Anesthesiology Clinic; Ali Yalcindag, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Biochemistry Clinic; Tuba Hanci, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Biochemistry Clinic; Haluk Gümüs, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Anesthesiology Clinic; Namik Delibas, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Biochemistry Clinic; Emel Gönen, Consultant, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Orthopedics Clinic
Locations (1):
- Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital Anesthesiology and Biochemistry Clinics, Ankara, Turkey (Türkiye)